CLINICAL TRIAL: NCT01969526
Title: Effectiveness of a Multifactorial Intervention to Modify Frailty Parameters in Elderly Population
Brief Title: Effectiveness of a Multifactorial Intervention on Frailty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI12/01503
Record Dates: First submitted 2013-08-01; First posted 2013-10-25 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-03

CONDITIONS: Frail Elderly; Cognitive Impairment; Dependence
Keywords: Frail elderly
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifactorial Intervention (Experimental): Intervention consists in three different actions on frailty dimensions, applied to each subject in the intervention group, in groups of 15 participants: rehabilitative therapy plus intake of hyperproteic shakes, memory workshop and review of the medication.
  Interventions: Other: Multifactorial intervention
- No intervention (No Intervention): Usual care

INTERVENTIONS:
Other: Multifactorial intervention — Intervention consists in three different actions on frailty dimensions, applied to each subject in the intervention group, in groups of 15 participants: rehabilitative therapy and physical exercise plus intake of hyperproteic shakes, memory workshop and review of the medication.
  Other Names: Multifactorial intervention on frailty dimensions
  Arms: Multifactorial Intervention

SUMMARY:
Objective: To evaluate the effectiveness of a multifactorial intervention program based on physical activity and diet, memory workshops and review of medication, to modify frailty parameters, muscle strength and physical and cognitive performance in people 65 years or older with a positive screening for frailty. Secondly, to assess changes in falls, hospitalizations, nutritional risk, disability and institutionalization or home-care.

Methods: randomized clinical trial with a control group, of one year and a half of follow-up, conducted in eight primary care teams in Barcelona. Individuals to be included are 65 years or older with positive frailty screening, timed get-up-and-go between 10 to 30 seconds, and cognitive Lobo test greater than or equal to 18. 165 patients will be selected in each group (difference to be detected on physical performance (Short physical performance battery (SPPB)): 0.5 units; common Standard Deviation : 1.42, 20% lost to follow-up).

Intervention: consists in three different actions on frailty dimensions, applied to each subject in the intervention group, in groups of 15 participants: rehabilitative therapy plus intake of hyperproteic shakes, memory workshop and review of the medication.

Evaluations will be blinded and conducted at 0, 3 and 18 months. Analysis of variance for repeated measures to adjust for differences attributable to intervention effect and for potential confounders such as comorbidity, sensory limitations, social risk, other medical or social interventions, among others.

ELIGIBILITY:
Inclusion Criteria:

* Positive Barber screen
* Timed get-up-and-go 10 to 20 seconds
* cognitive Lobo test greater than or equal to 18

Exclusion Criteria:

* Home Care
* Institutionalization
* Conditions not allowing physical exercise

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 352 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Short Physical performance battery at 3 and 18 months | 0,3,18 months
  The Short Physical Performance Battery (SPPB) is a standardised assessment tool of lower limb function, testing 3 dimensions: standing balance, walking speed, and chair stands. Each component is scored between 0-4, total score from 0 (poor performance) to 12 (best performance).
Change from Baseline in Muscle strength at 3 and 18 months | 0,3,18 months
  Evaluation of upper extremities strength was assessed through the measurement of force with a handgrip dynamometer. Grip strength was evaluated using a portable hand dynamometer (JAMAR®0-90 kg, coding 506320). The participants were seated with their shoulder in a neutral position and their elbow flexed at 90°. Three attempts were performed alternately in each hand; the mean of the three measures was recorded.
Change from Baseline in Cognitive Performance (Barcelona test) at 3 and 18 months | 0,3,18 months
  The first neuro-psychometric instrument developed in Spain to measure semi-quantitatively cognitive status in clinical neurology was the Barcelona Test (BT). Shortened version of the BT, named Barcelona Test Review (BTR) had been used for neuropsychological area evaluation in our participants and it takes only 20-30 minutes to administer

SECONDARY OUTCOMES:
Number of Participants with Falls during follow-up, at 18 months | 18 months
Change from Baseline in Functional Capacity at 18 months | 18 months
  Barthel Index Lawton&Brody Index
Number of Participants Hospitalized during follow-up, at 18 months | 18 months
Number of Participants Institutionalized during follow-up, at 18 months | 18 months
Number of Participants included in Home Health care during follow-up, at 18 months | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Josep Maria segura, MD, Phd, Principal Investigator — Jordi Gol Foundation
Locations (1):
- Institut Català de la Salut, Barcelona, Spain

REFERENCES:
- [Background] Romera L, Orfila F, Segura JM, Ramirez A, Moller M, Fabra ML, Lancho S, Bastida N, Foz G, Fabregat MA, Marti N, Cullell M, Martinez D, Gine M, Bistuer A, Cendros P, Perez E. Effectiveness of a primary care based multifactorial intervention to improve frailty parameters in the elderly: a randomised clinical trial: rationale and study design. BMC Geriatr. 2014 Nov 27;14:125. doi: 10.1186/1471-2318-14-125. PMID 25427568